CLINICAL TRIAL: NCT00380978
Title: Early Compared With Late Neuraxial Analgesia in Nulliparous Labor Induction
Brief Title: Neuraxial Versus Systemic Analgesia for Latent Phase Labor Effect on Rate of Operative Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: International Anesthesia Research Society (IARS) (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0524-009
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Labor Pain; Pregnancy
Keywords: labor pain; cesarean section; epidural analgesia; opioid analgesics; local anesthetics; labor induced
MeSH Terms: conditions — Labor Pain | interventions — Hydromorphone; Narcotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early analgesia:combined-spinal epidural (Active Comparator)
  Interventions: Procedure: combined spinal epidural analgesia
- late analgesia (systemic) (Active Comparator)
  Interventions: Procedure: late analgesia (systemic)

INTERVENTIONS:
Procedure: combined spinal epidural analgesia — Analgesia was initiated in the early group using a standard needle-through-needle technique with intrathecal fentanyl 25 mcg and an epidural test dose of lidocaine 15 mg/ml and epinephrine 5 mcg/ml in 3ml. At the second analgesia request, the cervix was examined. Epidural analgesia was initiated with a dilute bupivicaine/fentanyl solution if the cervix was less than 4 cm. If the cervix was 4 cm or more, epidural analgesia was initiated with bupivicaine 1.25 mg/ml. If no cervical exam was performed at the second request for analgesia, the cervix was assumed to be at least 4 cm dilated. Thereafter, analgesia was maintained in all participants in the early group with patient-controlled epidural analgesia.
  Other Names: CSE
  Arms: early analgesia:combined-spinal epidural
Procedure: late analgesia (systemic) — Analgesia was initiated in the late group with hydromorphone 1mg intramuscularly (IM) and 1 mg intravenously (IV). If the cervix was less than 4 cm at the second analgesia request, hydromorphone analgesia was repeated. Epidural analgesia was initiated with bupivicaine 1.25 mg/ml if the cervix was 4 cm or more. At the third analgesia request, epidural analgesia was initiated regardless of cervical dilation. Thereafter, epidural analgesia was maintained with patient controlled analgesia until delivery.
  Other Names: Dilaudid, narcotic
  Arms: late analgesia (systemic)

SUMMARY:
The purpose of this study in nulliparous women undergoing induction of labor is to determine whether initiation of neuraxial analgesia compared to systemic opioid analgesia early in labor (< 4 cm cervical dilation)affects the cesarean delivery rate.

DETAILED DESCRIPTION:
Women in early labor frequently request pain medication. Obstetricians may prescribe narcotics (administered as an intravenous (IV) or intramuscular (IM) injection). However, IV or IM narcotics provide incomplete pain relief and have maternal and fetal/neonatal side effects, e.g., maternal drowsiness, respiratory depression, nausea, vomiting, and neonatal respiratory depression. Other obstetricians allow their patients to request early neuraxial (spinal or epidural) analgesia. The results of several studies comparing patients who received epidural versus IV/IM narcotic labor analgesia (not specifically in early labor)suggest that initiation of early neuraxial analgesia may be associated with higher Cesarean delivery rates. It has been hypothesized that epidural/spinal local anesthetics may induce pelvic musculature relaxation leading to failure of fetal descent and rotation. However, early pain may be a marker for other factors that increase the risk of Cesarean delivery, e.g., large or malpositioned baby, or dysfunctional labor. Whether or not early neuraxial analgesia (particularly if narcotic based, which would not cause pelvic muscle paralysis) compared to IV/IM narcotics, adversely affects the outcome of labor has not been studied in a randomized, prospective fashion. The purpose of this study is to compare Cesarean and forcep delivery rates, and quality of pain relief, in first-time mothers undergoing induction of labor who receive neuraxial versus IV/IM analgesia for early labor (cervical dilation < 4 cm).

ELIGIBILITY:
Inclusion Criteria:

* induction of labor
* nulliparity
* >36 weeks gestation
* singleton
* vertex position
* cervical dilation < 4 cm at first request for analgesia
* desires neuraxial analgesia

Exclusion Criteria:

* spontaneously laboring
* multiparity
* nonvertex presentation
* at or >4cm at analgesia request
* chronic opioid therapy
* acute opioid therapy within 4 hours of analgesia request
* allergy to study drugs (hydromorphone, fentanyl, bupivacaine, lidocaine)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1026 (Actual)
Dates: Start 2001-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Wong CA, Scavone BM, Peaceman AM, McCarthy RJ, Sullivan JT, Diaz NT, Yaghmour E, Marcus RJ, Sherwani SS, Sproviero MT, Yilmaz M, Patel R, Robles C, Grouper S. The risk of cesarean delivery with neuraxial analgesia given early versus late in labor. N Engl J Med. 2005 Feb 17;352(7):655-65. doi: 10.1056/NEJMoa042573. PMID 15716559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2001 and December 2006, women presenting at Prentice Women's Hospital for induction of labor and who desired neuraxial analgesia were eligible to participate. Patients were asked to participate by study personnel after admission to the Labor and Delivery Unit and gave written informed consent before request for analgesia.
Pre-assignment Details: A total of 1,026 women consented to participate. 208 women were excluded because cervical dilation was 4 cm or more at the first analgesia request. Twelve participants were excluded after randomization because they did not receive the allocated intervention and outcome data were not available. The remaining 806 women were included in the analysis.
Groups:
- Early Analgesia:Combined-spinal Epidural: Laboring women with induction of labor requesting analgesia at cervical dilation less than 4 cm randomized to receive spinal fentanyl 25 micrograms and epidural bupivacaine 6.25 mg/ml and fentanyl 1.96 micrograms/ml for labor analgesia.
- Systemic Analgesia: Laboring women with induction of labor requesting analgesia at cervical dilation less than 4 cm randomized to receive hydromorphone 1mg IM and 1mg IV until cervical dilation greater than 4 cm or third request for analgesia. Epidural
Period: Overall Study
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Started | 408 | 410
Completed | 406 | 400
Not Completed | 2 | 10
Not completed — Refused allocated intervention | 0 | 6
Not completed — Wrong study envelope | 0 | 2
Not completed — Allocation prior to analgesia request | 1 | 2
Not completed — Parous patient | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia | Total
Number analyzed (Participants) | 408 | 410 | 818
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 408 | 410 | 818
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6) | 31 (5) | 31 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 408 | 410 | 818
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 408 | 410 | 818

OUTCOME MEASURES:

1. Primary Outcome: Delivered by Cesarean Section
Description: The decision to proceed to operative delivery was made by the obstetric team for maternal or fetal indications.
Time Frame: Time form initiation of labor analgesia to delivery (up to 24 hours)
Population: Analysis per protocol. 10 did not receive intervention in combined spinal epidural group and 2 in the systemic analgesia group
Measure: Number; unit: participants
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Number analyzed (Participants) | 406 | 400
participants | 134 | 126
Statistical Analysis 1: Comparison: Early Analgesia:Combined-spinal Epidural vs Systemic Analgesia; Group sample sizes of 800 in each group achieve 80% power to detect equivalence when the margin of equivalence extends from 0.1 to 0.25; Test type: Non-Inferiority or Equivalence — Equivalence; p = 0.65, Chi-squared, Corrected; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.90 to 1.20]

2. Secondary Outcome: Instrumented Vaginal Delivery
Description: The decision to proceed to assisted/instrumental delivery was made by the obstetric team for maternal or fetal indications.
Time Frame: At time of decision for delivery
Population: Per protocol - subjects that delivered vaginally
Measure: Number; unit: participants
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Number analyzed (Participants) | 272 | 274
participants | 57 | 59
Statistical Analysis 1: Comparison: Early Analgesia:Combined-spinal Epidural vs Systemic Analgesia; There rate of instrumented vaginal delivery will be equal in both groups; Test type: Superiority or Other; p = 0.63, Chi-squared; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.80 to 1.20]

3. Secondary Outcome: Duration of Labor
Description: Labor was induced by initiating an oxytocin infusion or by infusing extra-amniotic saline followed by oxytocin. All participants had continuous external electronic fetal heart rate (FHR) monitoring and tocodynamometry. Internal fetal scalp electrodes were placed when the external tracing was not interpretable, and intrauterine pressure catheters were used to measure the intensity of contractions when deemed necessary by the obstetricians. Artificial rupture of membranes was performed, and nurses titrated oxytocin infusions according to institutional protocol.
Time Frame: Initiation of induction of labor to time of delivery
Population: Per protocol
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Number analyzed (Participants) | 406 | 400
minutes | 528 [491 to 564] | 569 [538 to 600]
Statistical Analysis 1: Comparison: Early Analgesia:Combined-spinal Epidural vs Systemic Analgesia; Test type: Superiority or Other; p = 0.047, Log Rank

4. Secondary Outcome: Indication for Cesarean Delivery
Description: The decision to proceed to operative delivery was made by the obstetric team for maternal or fetal indications.
Time Frame: At time of decision for delivery
Population: Number of cesarean deliveries
Measure: Number; unit: participants
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Number analyzed (Participants) | 134 | 126
participants
  Arrested dilation | 85 | 83
  Arrested descent | 18 | 23
  Non-reassuring fetal status | 27 | 16
  Other | 4 | 4
Statistical Analysis 1: Comparison: Early Analgesia:Combined-spinal Epidural vs Systemic Analgesia; Test type: Superiority or Other; p = 0.35, Chi-squared

5. Secondary Outcome: Analgesia Efficacy
Description: Patients were asked to rate their average pain score using an 11-point verbal rating score (VRS)for pain (0 - 10: 0= no pain, 10= worst pain imaginable) between 1st and 2nd analgesia request.
Time Frame: At first and second analgesia requests
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Number analyzed (Participants) | 406 | 400
Scores on a scale | 1 [0 to 3] | 5 [3 to 6]
Statistical Analysis 1: Comparison: Early Analgesia:Combined-spinal Epidural vs Systemic Analgesia; Test type: Superiority or Other; p < 0.005, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -4, 95% CI 2-sided [-4 to -3]

6. Secondary Outcome: Nausea
Description: Participants were asked to rate their nausea (as none, mild, moderate, or severe) and report the presence or absence of vomiting.
Time Frame: At second analgesia request
Measure: Number; unit: participants
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Number analyzed (Participants) | 406 | 400
participants
  None | 372 | 265
  Mild | 25 | 69
  Moderate | 5 | 49
  Severe | 2 | 16
Statistical Analysis 1: Comparison: Early Analgesia:Combined-spinal Epidural vs Systemic Analgesia; Test type: Superiority or Other; p < 0.005, Chi-squared, Corrected

7. Secondary Outcome: Neonatal Outcome (APGAR Score < 7 at 5 Minutes)
Description: Infant's Apgar scores measured at 5 minutes of life and were assigned by nurses and pediatricians responsible for neonatal assessment. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing the five values. The categories are skin color, pulse, reflex to stimulation, muscle tome, and breathing. The test was done at one and five minutes after birth, and may be repeated later if the score is and remains low. Scores 3 and below are generally regarded as critically low, 4 to 6 fairly low, and 7 to 10 generally normal.
Time Frame: APGAR score at 5 minutes
Measure: Number; unit: participants
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Number analyzed (Participants) | 406 | 400
participants | 14 | 6
Statistical Analysis 1: Comparison: Early Analgesia:Combined-spinal Epidural vs Systemic Analgesia; Test type: Superiority or Other; p = 0.11, Fisher Exact

8. Secondary Outcome: Vomiting
Description: Vomiting during labor analgesia
Time Frame: Vomiting at second analgesia request
Measure: Number; unit: participants
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Number analyzed (Participants) | 406 | 400
participants | 12 | 61
Statistical Analysis 1: Comparison: Early Analgesia:Combined-spinal Epidural vs Systemic Analgesia; Test type: Superiority or Other; p < 0.005, Chi-squared, Corrected

ADVERSE EVENTS:
Arm/Group | Early Analgesia:Combined-spinal Epidural | Systemic Analgesia
Serious Adverse Events (participants affected / at risk) | 0/406 | 0/400
Other Adverse Events (participants affected / at risk) | 32/406 | 134/400
OTHER ADVERSE EVENTS (reported when occurring in more than 0.10% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Analgesia:Combined-spinal Epidural (N=406) | Systemic Analgesia (N=400)
Nausea and/or vomiting (Gastrointestinal disorders) | 32 (32) | 134 (134) — Patient self assessment of nausea and or vomiting following analgesia treatment. All subjects that vomited reported nausea prior to vomiting.

LIMITATIONS AND CAVEATS:
The study was not powered to detect a small difference between groups in the cesarean delivery rate. It was not blinded. Different obstetric providers have different management styles, and different triggers for performing cesarean delivery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes